CLINICAL TRIAL: NCT04869813
Title: Sarcopenia Characterization Using Magnetic Resonance Fingerprinting and Phosphorous Magnetic Resonance Spectroscopic Imaging Evaluation (SUSIE)
Brief Title: Sarcopenia Magnetic Resonance Imaging Evaluation (SUSIE)
Acronym: SUSIE
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wilson Tang, Staff Cardiovascular and Metabolic Sciences, The Cleveland Clinic
Other Study IDs: 21-124
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart failure patients: Inclusion criteria:
  * Age > or = 40 yrs
  * Stable chronic heart failure
  * Systolic dysfunction determined by cardiac MRI with left ventricle ejection fraction 40% or less
  Exclusion criteria:
  • Advanced liver disease, advanced cancer, advanced chronic obstructive pulmonary disease
  Contraindications to MRI such as:
  * Heart pacemaker/defibrillator
  * Electronic/implanted stimulators or devices, including deep brain stimulator, vagus nerve stimulator, bladder stimulator, spine stimulator, neurostimulators; implanted electrodes or wires
  * Cochlear implant or other ear implants
  * Implanted drug pumps (insulin, narcotic/pain medications, drugs to treat spasticity)
  * Programmable shunt
  * Aneurysm clips and coils
  * Stents • Filters (for example, blood clot filters)
  * Metal fragment in body or eye (eg, BBs, bullets, shrapnel, metal pieces or shavings)
- Healthy volunteers (Controls): Inclusion criteria:
  * Age > or = 40 yrs
  * No diagnosed heart failure or sarcopenia
  Exclusion criteria
  • Advanced liver disease, advanced cancer, advanced chronic obstructive pulmonary disease
  Contraindications to MRI such as:
  * Heart pacemaker/defibrillator
  * Electronic/implanted stimulators or devices, including deep brain stimulator, vagus nerve stimulator, bladder stimulator, spine stimulator, neurostimulators; implanted electrodes or wires
  * Cochlear implant or other ear implants
  * Implanted drug pumps (insulin, narcotic/pain medications, drugs to treat spasticity)
  * Programmable shunt
  * Aneurysm clips and coils
  * Stents
  * Filters (for example, blood clot filters)
  * Metal fragment in body or eye (eg, BBs, bullets, shrapnel, metal pieces or shavings)

SUMMARY:
The goal of the proposed research is to investigate Magnetic Resonance (MR) Fingerprinting and P-MRS (Phosphorus-31 MR Spectroscopy) imaging for characterization of skeletal muscle in heart failure patients with sarcopenia. Heart failure patients with and without sarcopenia will be scanned using MR Fingerprinting and an existing Post-exercise phosphocreatine (PCr) recovery MR imaging protocol to obtain characteristic profiles of quantitative T1, T2, and PCr recovery rate.

DETAILED DESCRIPTION:
Sarcopenia is a common comorbidity and predictor of mortality in heart failure that is characterized by a loss of muscle mass and functional strength. Sarcopenia, in heart failure and other chronic diseases, has been consistently predictive of poor outcomes. However, current tools to identify the presence of sarcopenia, such as functional tests and questionnaires are indirect, non-specific, and not effective until patients have reached an overtly cachectic state and significant muscle deterioration has already occurred. MRI can serve an important, noninvasive role in the assessment and management of sarcopenia by providing insight as to tissue microstructure and mitochondrial function. For example, MRI has shown significant changes in T2 relaxation time, diffusion fractional anisotropy, and lipid content in skeletal muscle of pre-frail/frail patients as compared to healthy volunteers. Post-exercise phosphocreatine (PCr) recovery, evaluated using phosphorus-31 (P) MR spectroscopy Imaging(P-MRSI), has shown impairment of mitochondrial function in pre-frail elderly as compared to active elderly. MR fingerprinting (MRF) is a promising tool for tissue characterization via rapid, robust quantification of T1 and T2 relaxation and has been shown to be accurate and reproducible across sites. Despite applications in neuroimaging and cardiac imaging, MRF has had limited use in musculoskeletal imaging and has not been investigated for use in characterizing sarcopenia. Similarly, P-MRS imaging has not been employed for evaluation of sarcopenia in heart failure patients, a population which may have a unique etiology from other sarcopenia phenotypes. Characterization of sarcopenia may support a range of rapidly developing treatment options in this population. While evidence suggests exercise therapy can improve frailty status, for instance in 39% of patients at 12 month follow-up, it is not yet well-understood which patients will respond to treatment. With a range of treatment options such as nutritional supplementation, hormone therapy, and cardiovascular drugs, MRF and P-MRSI could serve as powerful noninvasive tools to provide a personalized approach for sarcopenic phenotypes, match them to appropriate therapy, and monitor therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients

  * Age ≥40 yrs
  * Stable chronic heart failure
  * Systolic dysfunction determined by cardiac MRI with left ventricle ejection fraction 40% or less
* Healthy Volunteers

  * Age ≥40 yrs
  * No diagnosed heart failure or sarcopenia

Exclusion Criteria:

* Heart failure patients

  • Advanced liver disease, advanced cancer, advanced chronic obstructive pulmonary disease
* Healthy volunteers (controls)

  * Advanced liver disease, advanced cancer, advanced chronic obstructive pulmonary disease
  * Contraindications to MRI Contraindications to MRI
  * Heart pacemaker/defibrillator
  * Electronic/implanted stimulators or devices, including deep brain stimulator, vagus nerve stimulator, bladder stimulator, spine stimulator, neurostimulators; implanted electrodes or wires
  * Cochlear implant or other ear implants
  * Implanted drug pumps (insulin, narcotic/pain medications, drugs to treat spasticity)
  * Programmable shunt
  * Aneurysm clips and coils
  * Stents
  * Filters (for example, blood clot filters)
  * Metal fragment in body or eye (eg, BBs, bullets, shrapnel, metal pieces or shavings)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure and Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Anticipated Results | 3 years
  This proposal is expected to produce information as to the change in T1, T2, muscle area, fat fraction, and PCr recovery rate values for heart failure patients with sarcopenia as compared to non-sarcopenic volunteers. Future work will expand upon this study to evaluate to progression of sarcopenia, and evaluate the prognostic value of imaging biomarkers (T1, T2, muscle area, fat fraction, PCr recovery) in predicting heart failure and sarcopenic related outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: W. H. Wilson Tang, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States